CLINICAL TRIAL: NCT03866174
Title: A Randomized, Double-Blind, Support-of-Concept Phase 2 Study of Single-Dose Psilocybin for Major Depressive Disorder (MDD)
Brief Title: A Study of Psilocybin for Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Usona Institute (Other)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSIL201
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Depressive Disorder, Major
Keywords: Psilocybin, Psychedelics, Depression, MDD
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Psilocybin; Niacin; Niacinamide; SET protein, human; Clinical Protocols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin (Experimental): Participants will receive a single 25 mg dose of psilocybin along with the Set and Setting (SaS) protocol. Psilocybin is administered orally as a capsule and taken with water.
  Interventions: Drug: Psilocybin; Other: Set and Setting (SaS) Protocol
- Niacin (Active Comparator): Participants will receive a single 100 mg dose of niacin along with the Set and Setting (SaS) protocol. Niacin is administered orally as a capsule and taken with water.
  Interventions: Drug: Niacin; Other: Set and Setting (SaS) Protocol

INTERVENTIONS:
Drug: Psilocybin — The psilocybin used in this study is synthetically manufactured in a laboratory and meets quality specifications suitable for human research use. The active drug is encapsulated using a hydroxypropyl methylcellulose (HPMC) capsule and contains 25 mg of psilocybin.
  Other Names: Psilocybine, Psilocibin, Indocybin
  Arms: Psilocybin
Drug: Niacin — The active placebo is encapsulated using a HPMC capsule and contains 100 mg of pharmaceutical grade niacin.
  Other Names: Vitamin B3
  Arms: Niacin
Other: Set and Setting (SaS) Protocol — The SaS Protocol prescribes 6-8 hours of preparatory meetings with two facilitators prior to dosing, a 7-10 hour dosing session in a comfortable room under the supervision of the same two facilitators, and 4 hours of post-dose integration sessions with facilitators. During the dosing session participants are encouraged to wear eyeshades and listen to a curated playlist on headphones.

SUMMARY:
One hundred participants, ages 21 to 65, who meet Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for major depressive disorder (MDD) will be stratified by study site and randomized with a 1-to-1 allocation under double-blind conditions to receive a single 25 mg oral dose of psilocybin or a single 100 mg oral dose of niacin. Niacin will serve as an active placebo.

The purpose of this study is to evaluate the potential efficacy of a single 25 mg oral dose of psilocybin for MDD compared to the active placebo in otherwise medically-healthy participants, assessed as the difference between groups in changes in depressive symptoms from Baseline to Day 43 post-dose.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) has become a health crisis of epidemic proportions in the modern world. One in six individuals in the United States will experience an episode of major depression in his or her lifetime, and it is estimated that major depression will rank second after cardiac disease as a cause of international medical morbidity by the year 2020. Depression is associated with greater disability than are most other chronic illnesses and is a risk factor for mortality. Additionally, depression predicts the later development of a number of medical conditions, including cardiac and cerebrovascular disease, hypertension, diabetes, obesity, metabolic syndrome, dementia, and cancer. Unfortunately, most patients with depression do not experience a complete resolution of symptoms with antidepressant treatment. Partial-but incomplete-response to antidepressants is associated with an increased risk of full symptomatic relapse (even when on therapy) and a worse long-term disease course. Combined with the high prevalence and significant disability associated with MDD, the fact that currently available treatments are not fully adequate highlights the tremendous need to identify novel treatment strategies.

Data suggest that psilocybin may have behavioral effects relevant to the treatment of depression and recent studies also suggest that psilocybin may possess antidepressant properties. To further assess the effects of psilocybin on MDD signs and symptoms, this trial will enroll 100 participants, ages 21 to 65, who meet criteria for MDD. Participants will be stratified by study site and randomized with a 1-to-1 allocation under double-blind conditions to receive a single 25 mg oral dose of psilocybin or a single 100 mg oral dose of niacin. Niacin will serve as an active placebo.

To enhance participant safety, a Set and Setting (SaS) protocol will be utilized similar to the protocol that has been used in all modern studies of psilocybin. The SaS protocol for this study includes: 1) a period of preparation with session Facilitators prior to dosing; 2) administration of study medications in an aesthetically pleasing room under the supervision of two Facilitators who are present throughout the session; and 3) three post-dose integration sessions during which participants are encouraged to discuss their intervention experience with the Facilitators. The SaS protocol will be identical for those randomized to psilocybin or active placebo.

The primary objective of this study is to evaluate the potential efficacy of a single 25 mg oral dose of psilocybin for MDD compared to the active placebo (niacin), assessed as the difference between groups in changes in depressive symptoms from Baseline to Day 43 post-dose.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 65 years old
* Able to swallow capsules
* If of childbearing potential, agree to practice an effective means of birth control throughout the duration of the study
* Have an identified support person and agree to be accompanied home by that person following dosing
* Have sustained moderate-severe depression symptoms at Screening and Baseline
* Meet DSM-5 criteria for a diagnosis of major depressive disorder and are currently experiencing a major depressive episode of at least a 60-day duration at the time of screening

Exclusion Criteria:

* Women who are pregnant or who intend to become pregnant during the study or who are currently nursing
* Have any of the following cardiovascular conditions: uncontrolled hypertension, coronary artery disease, congenital long QT syndrome, cardiac hypertrophy, cardiac ischemia, congestive heart failure, myocardial infarction, tachycardia, artificial heart valve, a clinically significant screening ECG abnormality, or any other significant cardiovascular condition
* Have a history of stroke or Transient Ischemic Attack (TIA)
* Have moderate to severe hepatic impairment
* Have epilepsy
* Have insulin-dependent diabetes
* Have a positive urine drug test
* Nicotine dependence that would disallow an individual to be nicotine free for the 7-10 hours during the dosing period
* Meet DSM-5 criteria for schizophrenia spectrum or other psychotic disorders, including major depressive disorder with psychotic features, or Bipolar I or Bipolar II Disorder
* Meet DSM-5 criteria for antisocial personality disorder
* Meet DSM-5 criteria for a moderate or severe alcohol or drug use disorder

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Change in central rater Montgomery-Asberg Depression Rating Scale (MADRS) total score from Baseline to post-dose Day 43 | Baseline; Day 43 post-dose
  The MADRS is a clinician-rated scale designed to measure depression severity and to detect changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition. The total (composite) MADRS score is used as the endpoint.

SECONDARY OUTCOMES:
Change in central rater MADRS score from Baseline to post-dose Day 8 | Baseline, Day 8 post-dose
  The MADRS is a clinician-rated scale designed to measure depression severity and to detect changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition. The total (composite) MADRS score is used as the endpoint.
Change in on-site rater administered Sheehan Disability Scale (SDS) score from Baseline to post-dose Day 43 | Day 8, 15, 29, and 43 post-dose
  The SDS is a composite of three self-rated items designed to measure the extent to which three major sectors in the patient's life are impaired by psychiatric symptoms, including depression.
Sustained depressive symptom response defined as a ≥ 50% reduction from Baseline central rater MADRS score at all post-dose assessments | Day 8, 15, 29, and 43 post-dose
  The MADRS is a clinician-rated scale designed to measure depression severity and to detect changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition. The total (composite) MADRS score is used as the endpoint.
Sustained depressive symptom remission defined as a central rater MADRS total score ≤ 10 at all post-dose assessments | Day 8, 15, 29, and 43 post-dose
  The MADRS is a clinician-rated scale designed to measure depression severity and to detect changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition. The total (composite) MADRS score is used as the endpoint.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of California, San Francisco, San Francisco, California
  - Pacific Neuroscience Institute, Santa Monica, California
  - Yale University, New Haven, Connecticut
  - Segal Trials, Lauderhill, Florida
  - Emory University, Atlanta, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Hassman Research Institute, Berlin, New Jersey
  - New York University School of Medicine, New York, New York
  - Cedar Clinical Research, Draper, Utah
  - University of Wisconsin - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carhart-Harris RL, Leech R, Hellyer PJ, Shanahan M, Feilding A, Tagliazucchi E, Chialvo DR, Nutt D. The entropic brain: a theory of conscious states informed by neuroimaging research with psychedelic drugs. Front Hum Neurosci. 2014 Feb 3;8:20. doi: 10.3389/fnhum.2014.00020. eCollection 2014. PMID 24550805
- [Background] Nichols DE. Hallucinogens. Pharmacol Ther. 2004 Feb;101(2):131-81. doi: 10.1016/j.pharmthera.2003.11.002. PMID 14761703
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE, Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. doi: 10.1001/jama.289.23.3095. PMID 12813115
- [Background] Global Burden of Disease Study 2013 Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 301 acute and chronic diseases and injuries in 188 countries, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Aug 22;386(9995):743-800. doi: 10.1016/S0140-6736(15)60692-4. Epub 2015 Jun 7. PMID 26063472
- [Background] Wulsin LR, Vaillant GE, Wells VE. A systematic review of the mortality of depression. Psychosom Med. 1999 Jan-Feb;61(1):6-17. doi: 10.1097/00006842-199901000-00003. PMID 10024062
- [Background] Joynt KE, Whellan DJ, O'Connor CM. Depression and cardiovascular disease: mechanisms of interaction. Biol Psychiatry. 2003 Aug 1;54(3):248-61. doi: 10.1016/s0006-3223(03)00568-7. PMID 12893101
- [Background] Thomas AJ, Kalaria RN, O'Brien JT. Depression and vascular disease: what is the relationship? J Affect Disord. 2004 Apr;79(1-3):81-95. doi: 10.1016/S0165-0327(02)00349-X. PMID 15023483
- [Background] Davidson K, Jonas BS, Dixon KE, Markovitz JH. Do depression symptoms predict early hypertension incidence in young adults in the CARDIA study? Coronary Artery Risk Development in Young Adults. Arch Intern Med. 2000 May 22;160(10):1495-500. doi: 10.1001/archinte.160.10.1495. PMID 10826464
- [Background] Jonas BS, Lando JF. Negative affect as a prospective risk factor for hypertension. Psychosom Med. 2000 Mar-Apr;62(2):188-96. doi: 10.1097/00006842-200003000-00006. PMID 10772396
- [Background] Eaton WW, Armenian H, Gallo J, Pratt L, Ford DE. Depression and risk for onset of type II diabetes. A prospective population-based study. Diabetes Care. 1996 Oct;19(10):1097-102. doi: 10.2337/diacare.19.10.1097. PMID 8886555
- [Background] Kawakami N, Takatsuka N, Shimizu H, Ishibashi H. Depressive symptoms and occurrence of type 2 diabetes among Japanese men. Diabetes Care. 1999 Jul;22(7):1071-6. doi: 10.2337/diacare.22.7.1071. PMID 10388970
- [Background] Barefoot JC, Heitmann BL, Helms MJ, Williams RB, Surwit RS, Siegler IC. Symptoms of depression and changes in body weight from adolescence to mid-life. Int J Obes Relat Metab Disord. 1998 Jul;22(7):688-94. doi: 10.1038/sj.ijo.0800647. PMID 9705031
- [Background] Pine DS, Goldstein RB, Wolk S, Weissman MM. The association between childhood depression and adulthood body mass index. Pediatrics. 2001 May;107(5):1049-56. doi: 10.1542/peds.107.5.1049. PMID 11331685
- [Background] Raikkonen K, Matthews KA, Kuller LH. The relationship between psychological risk attributes and the metabolic syndrome in healthy women: antecedent or consequence? Metabolism. 2002 Dec;51(12):1573-7. doi: 10.1053/meta.2002.36301. PMID 12489070
- [Background] Jorm AF. History of depression as a risk factor for dementia: an updated review. Aust N Z J Psychiatry. 2001 Dec;35(6):776-81. doi: 10.1046/j.1440-1614.2001.00967.x. PMID 11990888
- [Background] Spiegel D, Giese-Davis J. Depression and cancer: mechanisms and disease progression. Biol Psychiatry. 2003 Aug 1;54(3):269-82. doi: 10.1016/s0006-3223(03)00566-3. PMID 12893103
- [Background] Greden JF. The burden of disease for treatment-resistant depression. J Clin Psychiatry. 2001;62 Suppl 16:26-31. PMID 11480881
- [Background] Judd LL, Akiskal HS, Maser JD, Zeller PJ, Endicott J, Coryell W, Paulus MP, Kunovac JL, Leon AC, Mueller TI, Rice JA, Keller MB. A prospective 12-year study of subsyndromal and syndromal depressive symptoms in unipolar major depressive disorders. Arch Gen Psychiatry. 1998 Aug;55(8):694-700. doi: 10.1001/archpsyc.55.8.694. PMID 9707379
- [Background] Miller IW, Keitner GI, Schatzberg AF, Klein DN, Thase ME, Rush AJ, Markowitz JC, Schlager DS, Kornstein SG, Davis SM, Harrison WM, Keller MB. The treatment of chronic depression, part 3: psychosocial functioning before and after treatment with sertraline or imipramine. J Clin Psychiatry. 1998 Nov;59(11):608-19. doi: 10.4088/jcp.v59n1108. PMID 9862607
- [Background] Simon GE. Long-term prognosis of depression in primary care. Bull World Health Organ. 2000;78(4):439-45. PMID 10885162
- [Background] Carhart-Harris RL, Bolstridge M, Rucker J, Day CM, Erritzoe D, Kaelen M, Bloomfield M, Rickard JA, Forbes B, Feilding A, Taylor D, Pilling S, Curran VH, Nutt DJ. Psilocybin with psychological support for treatment-resistant depression: an open-label feasibility study. Lancet Psychiatry. 2016 Jul;3(7):619-27. doi: 10.1016/S2215-0366(16)30065-7. Epub 2016 May 17. PMID 27210031
- [Background] Griffiths RR, Johnson MW, Carducci MA, Umbricht A, Richards WA, Richards BD, Cosimano MP, Klinedinst MA. Psilocybin produces substantial and sustained decreases in depression and anxiety in patients with life-threatening cancer: A randomized double-blind trial. J Psychopharmacol. 2016 Dec;30(12):1181-1197. doi: 10.1177/0269881116675513. PMID 27909165
- [Background] Ross S, Bossis A, Guss J, Agin-Liebes G, Malone T, Cohen B, Mennenga SE, Belser A, Kalliontzi K, Babb J, Su Z, Corby P, Schmidt BL. Rapid and sustained symptom reduction following psilocybin treatment for anxiety and depression in patients with life-threatening cancer: a randomized controlled trial. J Psychopharmacol. 2016 Dec;30(12):1165-1180. doi: 10.1177/0269881116675512. PMID 27909164
- [Derived] Raison CL, Sanacora G, Woolley J, Heinzerling K, Dunlop BW, Brown RT, Kakar R, Hassman M, Trivedi RP, Robison R, Gukasyan N, Nayak SM, Hu X, O'Donnell KC, Kelmendi B, Sloshower J, Penn AD, Bradley E, Kelly DF, Mletzko T, Nicholas CR, Hutson PR, Tarpley G, Utzinger M, Lenoch K, Warchol K, Gapasin T, Davis MC, Nelson-Douthit C, Wilson S, Brown C, Linton W, Ross S, Griffiths RR. Single-Dose Psilocybin Treatment for Major Depressive Disorder: A Randomized Clinical Trial. JAMA. 2023 Sep 5;330(9):843-853. doi: 10.1001/jama.2023.14530. PMID 37651119
- [Derived] Penn A, Dorsen CG, Hope S, Rosa WE. Psychedelic-Assisted Therapy: Emerging Treatments in Mental Health Disorders. Am J Nurs. 2021 Jun 1;121(6):34-40. doi: 10.1097/01.NAJ.0000753464.35523.29. PMID 33993135
- [Derived] Greenway KT, Garel N, Goyette N, Turecki G, Richard-Devantoy S. Adjunctive music improves the tolerability of intravenous ketamine for bipolar depression. Int Clin Psychopharmacol. 2021 Jul 1;36(4):218-220. doi: 10.1097/YIC.0000000000000363. PMID 33902087
- See also: World Health Organization Overview of Depression — http://www.who.int/mediacentre/factsheets/fs369/en/